CLINICAL TRIAL: NCT07174440
Title: Erector Spinae Plane Block in Patients Undergoing Lumbar Spine Fusion Surgery: Iohexol Spread, Extent of Block and Efficacy
Brief Title: Contrast and Anesthetic Level With Lumbar Erector Spinae Plan (ESP) Block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Salim M Hayek, Professor and Vice Chair for Clinical Research, Department of Anesthesiology, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20241500
Record Dates: First submitted 2025-09-12; First posted 2025-09-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pain
Keywords: Spinal surgery; ESP block
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Analgesia, Epidural; Dexmedetomidine; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spinal Surgery Participants (Experimental): Participants scheduled for spinal surgery will have ESP block medications administered as per standard care along with contrast dye.
  Interventions: Drug: Ropivacaine (Epidural analgesia); Drug: Dexmedetomidine; Drug: Iohexol; Procedure: QST Procedure

INTERVENTIONS:
Drug: Ropivacaine (Epidural analgesia) — The block solution will consist of 1% ropivacaine 3 mg/Kg ideal body weight (IBW) mixed with dexmedetomidine 0.5 mcg/Kg IBW and diluted with 10 mL iohexol 300 mg/mL and normal saline for a total volume of 40 mL. All medications used are standard of care
Drug: Dexmedetomidine — The block solution will consist of 1% ropivacaine 3 mg/Kg ideal body weight (IBW) mixed with dexmedetomidine 0.5 mcg/Kg IBW and diluted with 10 mL iohexol 300 mg/mL and normal saline for a total volume of 40 mL. All medications used are standard of care
Drug: Iohexol — The block solution will consist of 1% ropivacaine 3 mg/Kg ideal body weight (IBW) mixed with dexmedetomidine 0.5 mcg/Kg IBW and diluted with 10 mL iohexol 300 mg/mL and normal saline for a total volume of 40 mL. All medications used are standard of care except for iohexol which is used for study purposes.
Procedure: QST Procedure — The QST procedure (test of buzzing sensation and temperature sensation through pads applied to your skin) to assess the numb areas.

SUMMARY:
As per usual care for spine surgery, participants will have their back cleaned with alcohol and a needle will be placed using ultrasound for the ESP block. Through the needle, a small catheter will be placed in the participants back and the needle removed. Approximately one hour prior to the start of surgery, a numbing medication (ropivacaine, similar to Novocaine) in combination with dexmedetomidine (a pain medicine that is used in nerve block and that is not a narcotic) and contrast dye (iohexol) will be injected through the catheter. Participants will then go through the QST procedure (test of buzzing sensation and temperature sensation through pads applied to their skin) to assess the numb areas and then head to the operating room. In the operating room, the catheter will be removed after the surgeon obtains baseline CT scan images of the spine. Once surgery is completed, investigators will record pain scores over the next four days in the hospital and the amount of pain medication needed for controlling pain related to the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Adult patients 21-75 years of age
* ASA status: I-III
* Planned lumbar spine fusion involving no more than three levels
* Ability to ambulate prior to surgery

Exclusion Criteria:

* Previous lumbar spine surgery
* Metastatic cancer with involvement of the lumbar spine
* eGFR < 60 mL/min/1.73m2
* Active liver disease (hepatitis or cirrhosis)
* Confirmed allergy to ropivacaine, dexmedetomidine or iohexol
* Cognitive impairment resulting in inability to rate pain scores
* Patients receiving 30 mg or more of morphine equivalent daily dosing preoperatively
* Pregnancy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Verbal pain score as measured by the numerical rating scale (NRS) | 12 hours after surgery
  NRS rates pain intensity on a scale of 0 to 10, with 0 being no pain and 10 being worst possible pain.

SECONDARY OUTCOMES:
Patient-reported outcome to assess the quality of recovery as measured by the QoR-15 | Daily during hospital stay, up to 4 days
  Concise, 15-item questionnaire that covers domains like physical comfort, emotional state, psychological support, physical independence, and pain. A higher QoR-15 score indicates a better quality of recovery.
Time to oral food intake as measured by patient report | Daily during hospital stay, up to 4 days
Time to ambulation as measured by patient report | Daily during hospital stay, up to 4 days.
  Patients will be asked daily if they are walking to the bathroom.
Length of hospital stay as measured by medical record review | Up to 5 days
Number of intraoperative events as measured by medical record review. | Up to 12 hours after surgery
  Events include: hypotension, tachycardia, need for additional opioids beyond the study limit, and blood loss.

CONTACTS AND LOCATIONS:
Overall Officials: Salim Hayek, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No